CLINICAL TRIAL: NCT01437670
Title: A Prospective, Multicenter, Observation Study to Estimate the Dry Mouth in OAB Patients With Solifenacin
Brief Title: Observational Study to Estimate the Dry Mouth in OAB Patients With Solifenacin
Acronym: OAB
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); The Catholic University of Korea (Other); Ajou University (Other); Severance Hospital (Other); Cheil General Hospital and Women's Healthcare Center (Other); SMG-SNU Boramae Medical Center (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Myung-Soo Choo, Professor, Asan Medical Center
Other Study IDs: AMC 2011-0585
Record Dates: First submitted 2011-09-20; First posted 2011-09-21 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- dry mouth patients with solifenacin: dry mouth patients with solifenacin 5mg, 10mg
  Interventions: Drug: solifenacin 5mg, 10mg

INTERVENTIONS:
Drug: solifenacin 5mg, 10mg — solifenacin 5mg, 10mg
  Other Names: Vesicare

SUMMARY:
A prospective, multicenter, observation study to estimate the dry mouth in OAB patients with solifenacin

DETAILED DESCRIPTION:
To estimate the dry mouth and their impact on the efficacy of the drug in overactive bladder patients with solifenacin

ELIGIBILITY:
Inclusion Criteria:

* 1) male or female patients with 20 years of age or older 2) clinical history of OAB for at least 3 months prior to visit 2 3) more than 3 in total score and 2 in Q 3 index from OABSS questionnaire

Exclusion Criteria:

* 1) In clinical trial, female with pregnant, intent to become pregnant or breast-feeding 2)post-voided residual urine volume > 150ml 3) a history of catheterization due to acute urinary retention 4) a history of pelvic surgery within 6 months 5) 6) 7) a history of neurovascular disease such as Parkinson's disease, cerebral vascular disease, spinal injury or multiple sclerosis 8)patients with indwelling catheter or intermittent catheterization 9) active or recurrent (>3 episodes per year) urinary tract infection 10) the use of the following medication at least 2 weeks
* anticholinergics
* Tricyclic antidepressants,anti-epilepsy drug, anti-Parkinson's disease drug, anti-arrythmia drug type I
* Chlorpromazine, Thioridazine, Piperazine
* MAO inhibitor 11) Patient is currently taking or has taken within the past 4 weeks alpha-blocker for the treatment of benign prostatic hypertrophy 12) Patient is currently taking or has taken within the past 8 weeks 5ARI or estrogen medication 13) Patient is currently using or has used medications with known activities as inhibitors or inducers of cytochrome P4503A4 (CYP3A4)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with overactive bladder
  1. male or female patients with 20 years of age or older
  2. clinical history of OAB for at least 3 months prior to visit 2
  3. more than 3 in total score and 2 in Q 3 index from OABSS questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The changes of the total score in Xerostomia inventory XI from baseline | after 8 weeks of treatment from baseline
  11-item summated rating scale. Respondents were asked to choose one of five responses ('never', scoring 1~'very often', 5) total best and worst values: 11 and 49

SECONDARY OUTCOMES:
Global response assessment | after 8 weeks of treatment from baseline
  range, 1~7
The changes of the total score in overactive bladder symptom score (OABSS) from baseline | after 8 weeks treatment from baseline
  total best and worst values: 0 and 15
Visual Analog Scale (VAS) of dry mouth | after 8 weeks treatment from baseline
  The changes of the Visual Analog Scale (VAS) of dry mouth from baseline (range, 0~10)

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-Soo Choo, M.D., pH.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea